CLINICAL TRIAL: NCT01044251
Title: Frovatriptan as a Transitional Therapy in Medication Overuse Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Farnaz Amoozegar, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22522
Record Dates: First submitted 2010-01-05; First posted 2010-01-07 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Medication Overuse Headache; Analgesic Overuse Headache
Keywords: Medication overuse headache; Rebound headache; Analgesic overuse headache; Transitional therapy; Frovatriptan; Migraine
MeSH Terms: conditions — Headache Disorders, Secondary; Migraine Disorders | interventions — frovatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 10 days of treatment with placebo in a bid fashion that will look like the study medication.
  Interventions: Drug: Placebo
- Frovatriptan (Experimental): Frovatriptan 2.5 mg po bid for 10 days
  Interventions: Drug: Frovatriptan

INTERVENTIONS:
Drug: Frovatriptan — 2.5 mg po bid for 10 days
  Arms: Frovatriptan
Drug: Placebo — 1 tab po bid for 10 days
  Arms: Placebo

SUMMARY:
This study will analyze the effectiveness of a medication called Frovatriptan, in the context of medication overuse headache (MOH). MOH is a headache that develops when pain-killers are taken frequently. The treatment is to stop the overuse of these pain-killers, but that can sometimes worsen the headache first before it gets better. We are testing Frovatriptan against placebo to see if it can help patients with this transition and avoid the worsening of the headache that can occur. We will also see if Frovatriptan can help in other ways, such as maintain patients free of medication overuse.

DETAILED DESCRIPTION:
A single-centre, randomized, placebo-controlled trial is proposed to assess Frovatriptan as a transitional therapy in patients diagnosed with medication overuse headache. Currently, there are no proven transitional therapies to help patients get through the detoxification process. Frovatriptan has not been tested as a transitional therapy in the past. This study will compare Frovatriptan, taken over a 10 day transitional period, to placebo. The primary outcome of the study will be the mean headache intensity in the 10 day transitional period in the Frovatriptan group as compared to the placebo group. A number of secondary and exploratory outcomes will also be determined and further data collection will occur at 1, 2, and 3 month periods. The duration of the study for the participants will be 3 months, and they will be asked to keep detailed headache diaries during this time. Ten days of baseline headache diaries will also be performed before patients can enter the study.

ELIGIBILITY:
Inclusion Criteria:

* MOH diagnosed by IHS criteria
* Diagnosis of migraine (with or without aura) in past by IHS criteria
* If patients do not have a baseline diary, then a prospective diary for a 10-day period will be done to confirm medication overuse before study entry.
* Patients aged 18 to 65 years.
* Normal neurological examination.
* Patient is willing and able (in terms of capacity) to sign informed consent.
* Patient is able to understand and complete study protocol, including completion of headache diaries.
* Patient has a stable medical condition.

Exclusion Criteria:

* Headache not meeting IHS criteria for MOH.
* Presence of hemiplegic, basilar, ophthalmoplegic migraine or migrainous infarction.
* Findings on history, neurological exam, or neuroimaging suggestive of secondary causes of headache.
* Post-whiplash or post-traumatic headaches.
* Contraindications to triptans (such as heart disease, peripheral vascular disease or uncontrolled hypertension) or previous serious side effects/intolerance.
* Major psychiatric conditions (such as major depression, bipolar disorder, schizophrenia, addiction), either diagnosed by a physician or positive on standard clinic assessment tools (e.g. BDI questionnaire).
* Major medical conditions or treatments that may interfere with the patient's ability to participate in the study, such as dementia, advanced or terminal cancer, chemotherapy, etc.
* Patient is pregnant, breastfeeding, or is expecting to conceive within the time period of the study. Pregnancy will be determined using a urine test.
* Women of childbearing potential who are not using a reliable method of contraception.
* Patient is a recent user of illicit/recreational drugs or plans to use illicit drugs during the study time period.
* Patient has a recent history of alcohol abuse or dependence, or plans to abuse alcohol during the study duration.
* Patient is unlikely to comply with the study protocol, keep diaries and appointments, or does not have a fixed telephone or address.
* Patient is enrolled in another study or trial that may interfere with their participation or the results of this study.
* Patients with greater than 30% of their data missing during the ten days of baseline diary data collection.
* Patients with mean headache intensities of less than 3 (from a pain scale of 0 to 10, where 0=no pain and 10=pain as bad as possible) during the 10-day baseline period.
* Patients with ongoing Botox treatments or those who have received Botox in the last 4 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-01; Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
The mean headache intensity in the 10 day transitional period in the Frovatriptan group as compared to the placebo group. | After 10 days of therapy

SECONDARY OUTCOMES:
The difference in mean headache intensity between the 10 day transitional period and the baseline period. | After 10 days of therapy
The number of day segments with headache of grade 6 or higher during the 10 day transitional period and during days 11-20 of the study. | After 10 days and after 20 days
Number of headache-free days (grade zero) for first two months of study. | After 2 months
Proportion of patients free of medication overuse for first two months of study (i.e. less than 15 days of simple analgesic use or less than 10 days of other analgesic use per month). | After 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Werner J Becker, MD, FRCPC, Study Director — University of Calgary; Farnaz Amoozegar, MD, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- South Health Campus, Calgary, Alberta, Canada

REFERENCES:
- [Background] Grazzi L, Andrasik F, Usai S, Bussone G. Headache with medication overuse: treatment strategies and proposals of relapse prevention. Neurol Sci. 2008 Apr;29(2):93-8. doi: 10.1007/s10072-008-0867-8. Epub 2008 May 16. PMID 18483706
- [Background] Hagen K, Albretsen C, Vilming ST, Salvesen R, Gronning M, Helde G, Gravdahl G, Zwart JA, Stovner LJ. Management of medication overuse headache: 1-year randomized multicentre open-label trial. Cephalalgia. 2009 Feb;29(2):221-32. doi: 10.1111/j.1468-2982.2008.01711.x. Epub 2008 Sep 24. PMID 18823363
- [Background] Kelman L. Review of frovatriptan in the treatment of migraine. Neuropsychiatr Dis Treat. 2008 Feb;4(1):49-54. doi: 10.2147/ndt.s1871. PMID 18728819
- [Background] Markus F, Mikko K. Frovatriptan review. Expert Opin Pharmacother. 2007 Dec;8(17):3029-33. doi: 10.1517/14656566.8.17.3029. PMID 18001261